CLINICAL TRIAL: NCT05299346
Title: Post-ICU Covid19 Follow-up With Regards to Lung, Heart, Kidney and Cognitive Function
Brief Title: Post-ICU Follow-up Study in Covid-19 Patients
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgård, MD PhD Associate Professor, Sahlgrenska University Hospital
Other Study IDs: PICU COVID19
Record Dates: First submitted 2021-10-21; First posted 2022-03-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Pandemic; Intensive Care Unit Syndrome; Delirium
Keywords: covid19; Heart function; Lung function; Cognitive function
MeSH Terms: conditions — COVID-19; Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Post ICU covid survivors: Patients having survived and discharged from ICU care as a result of Covid 19
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — Comprehensive follow up in dedicated follow up unit

SUMMARY:
A follow up study of adult patients who have been treated in the ICU at Mölndal hospital due to Covid19 in the period of 2020 to 2022.

DETAILED DESCRIPTION:
The spread of Covid19 in the population in Sweden from 2019 and onwards posed new and serious strain on our ICU capacity. The disease presented with initially influenza like symptoms and evolved into multiorgan failure. 5% of all patients with verified Covid 19 were in need of critical care and among them the in-hospital mortality rate was 20%.

Patients will be followed up with after a minimum of three months after discharge from the ICU with regards to organ function.

Examinations within the scope of the study are;

* Comprehensive heart investigation including ultrasound
* Arterial blood gas and lung function tests including computer tomography of the lungs.
* Cognitive function with validated questioners
* Standardized test of physical function
* A panel of blood samples to assess organ function

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at the Intensive Care Unit at Mölndals hospital from 2020 to 2022 for Covid19
* More than 3 months passed since ICU discharge
* Over 18 years of age at time of inclusion
* Swedish resident with Swedish unique personal identification number.
* Informed consent

Exclusion Criteria:

* Under 18 years of age at time of inclusion
* Not a Swedish resident
* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that have been treated for Covid 19 at the ICU at Mölndal are eligible for participation
Sampling Method: Non-Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Lung Function oxygen saturation | One year
  Respiratory function following Covid19, saturation in SaO2%
Lung Function, end tidal Co2 in kPa | One year
  Respiratory function following Covid19, end tidal carbon dioxide in kPa,
Lung Function, complete arterial and venous blood gas in kPa | One year
  Respiratory function with arterial and venous blood gas pO2 and pCO2 in kPa
Lung Function spirometry | One year
  Respiratory function with spirometry in Volumes in ml related to BMI
Lung parenchym status | One year
  Ct scan of the lungs, assessed by radiology specialist, assessed for fibrosis, bronchiectasia and residual ground glass abnormalities
ECG | One year
  5 lead ECG for the detection av arrythmia
Cardiac ultrasound | One year
  Cardiac ultrasound including ejection fractions (EF%)
Cardiac biomarkers Troponin in ng/L | One year
  Cardiac function Blood sampling
Cardiac biomarkers NTproBNPin ng/L | One year
  Cardiac function Blood sampling
Cognitive function MMSE | One year
  Standardized cognitive tests
Cognitive function CDR | One year
  Standardized cognitive tests,
Cognitive function Montreal Cognitive Assessment | One year
  Standardized cognitive tests
Cognitive function biochemical markers | One year
  blood sampling with NFL, NSE, s-100B, fosfor-tau and APOE
Physical function | One year
  Standardized aggregate test of physical function, including seat raise test and grip strength measurement with validated instruments
Coagulation Status | One year
  Blood sampling Fibrinogen, D-Dimer, Antithrombin III and platelets, Aggregate variable to determine overall coagulation status
Covid 19 antibodies | One year
  Antibodies IgG against Covid 19 lab test

SECONDARY OUTCOMES:
Return to work | One year
  Are the subjects working or at the disposal of the labour market
Return to own home | one year
  Are the subjects living in their original housing or equivalent?
New need for nursing assistance at home? | one year
  Are the subjects in need of in home nursing care
Frailty | One year
  assessed accordingly to Clinical frailty scale
Mental fatigue | One Year
  self-assessment questionnaire Mental fatigue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to small sample size, anonymity will be difficult if data is shared

REFERENCES:
- [Background] Mahase E. Coronavirus covid-19 has killed more people than SARS and MERS combined, despite lower case fatality rate. BMJ. 2020 Feb 18;368:m641. doi: 10.1136/bmj.m641. No abstract available. PMID 32071063
- [Background] Pan XW, Xu D, Zhang H, Zhou W, Wang LH, Cui XG. Identification of a potential mechanism of acute kidney injury during the COVID-19 outbreak: a study based on single-cell transcriptome analysis. Intensive Care Med. 2020 Jun;46(6):1114-1116. doi: 10.1007/s00134-020-06026-1. Epub 2020 Mar 31. No abstract available. PMID 32236644
- [Background] Li XC, Zhang J, Zhuo JL. The vasoprotective axes of the renin-angiotensin system: Physiological relevance and therapeutic implications in cardiovascular, hypertensive and kidney diseases. Pharmacol Res. 2017 Nov;125(Pt A):21-38. doi: 10.1016/j.phrs.2017.06.005. Epub 2017 Jun 12. PMID 28619367
- [Background] Ronco C, Reis T. Kidney involvement in COVID-19 and rationale for extracorporeal therapies. Nat Rev Nephrol. 2020 Jun;16(6):308-310. doi: 10.1038/s41581-020-0284-7. PMID 32273593
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Wynants L, Van Calster B, Collins GS, Riley RD, Heinze G, Schuit E, Bonten MMJ, Dahly DL, Damen JAA, Debray TPA, de Jong VMT, De Vos M, Dhiman P, Haller MC, Harhay MO, Henckaerts L, Heus P, Kammer M, Kreuzberger N, Lohmann A, Luijken K, Ma J, Martin GP, McLernon DJ, Andaur Navarro CL, Reitsma JB, Sergeant JC, Shi C, Skoetz N, Smits LJM, Snell KIE, Sperrin M, Spijker R, Steyerberg EW, Takada T, Tzoulaki I, van Kuijk SMJ, van Bussel B, van der Horst ICC, van Royen FS, Verbakel JY, Wallisch C, Wilkinson J, Wolff R, Hooft L, Moons KGM, van Smeden M. Prediction models for diagnosis and prognosis of covid-19: systematic review and critical appraisal. BMJ. 2020 Apr 7;369:m1328. doi: 10.1136/bmj.m1328. PMID 32265220
- [Background] Terpos E, Ntanasis-Stathopoulos I, Elalamy I, Kastritis E, Sergentanis TN, Politou M, Psaltopoulou T, Gerotziafas G, Dimopoulos MA. Hematological findings and complications of COVID-19. Am J Hematol. 2020 Jul;95(7):834-847. doi: 10.1002/ajh.25829. Epub 2020 May 23. PMID 32282949
- [Background] Orde SR, Pulido JN, Masaki M, Gillespie S, Spoon JN, Kane GC, Oh JK. Outcome prediction in sepsis: speckle tracking echocardiography based assessment of myocardial function. Crit Care. 2014 Jul 11;18(4):R149. doi: 10.1186/cc13987. PMID 25015102
- [Background] Dalla K, Hallman C, Bech-Hanssen O, Haney M, Ricksten SE. Strain echocardiography identifies impaired longitudinal systolic function in patients with septic shock and preserved ejection fraction. Cardiovasc Ultrasound. 2015 Jul 2;13:30. doi: 10.1186/s12947-015-0025-4. PMID 26134971
- [Background] Dalla K, Bech-Hanssen O, Ricksten SE. Impact of norepinephrine on right ventricular afterload and function in septic shock-a strain echocardiography study. Acta Anaesthesiol Scand. 2019 Nov;63(10):1337-1345. doi: 10.1111/aas.13454. Epub 2019 Aug 19. PMID 31361336
- [Background] Rello J, Storti E, Belliato M, Serrano R. Clinical phenotypes of SARS-CoV-2: implications for clinicians and researchers. Eur Respir J. 2020 May 21;55(5):2001028. doi: 10.1183/13993003.01028-2020. Print 2020 May. PMID 32341111